CLINICAL TRIAL: NCT06804733
Title: Telemedicine-based Individualized Aerobic Exercise Training in Adults With Inactive or Mildly Active Inflammatory Bowel Disease: A Semi-crossover Randomized Controlled Trial
Brief Title: Efficacy of Individualized Aerobic Exercise Training in Patients With Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY2024SL379-01
Record Dates: First submitted 2024-12-27; First posted 2025-02-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week control intervention followed by 12-week aerobic exercise training (Active Comparator)
  Interventions: Behavioral: 12-week control intervention followed by 12-week aerobic exercise training
- 12-week aerobic exercise training directly (Experimental)
  Interventions: Behavioral: 12-week individualized aerobic exercise training

INTERVENTIONS:
Behavioral: 12-week individualized aerobic exercise training — After enrollment, subjects directly participate in a 12-week aerobic exercise training program. The training plan provides individualized progressive aerobic training based on their baseline physical activity level measured by International Physical Activity Questionnaire (IPAQ), with the exercise intensity being increased every four weeks.
  Arms: 12-week aerobic exercise training directly
Behavioral: 12-week control intervention followed by 12-week aerobic exercise training — After enrollment, subjects first undergo a 12-week control intervention (i.e., routine treatment) and then participate in a 12-week aerobic exercise training program. The training plan provides individualized progressive aerobic training based on their baseline physical activity level IPAQ, with the exercise intensity being increased every four weeks.
  Arms: 12-week control intervention followed by 12-week aerobic exercise training

SUMMARY:
The goal of this clinical trial is to learn if a 12-week individualized aerobic training program helps manage inactive or mildly active inflammatory bowel disease (IBD) including Crohn's disease (CD) and ulcerative colitis (UC) in adult patients aged 18-65 years. It will also assess participant compliance and the safety of the training program. The main questions it aims to answer are:

1. Does this aerobic training program improve the cardiopulmonary function of participants?
2. Does this aerobic training program help control disease activity?
3. Does this aerobic training program improve participants' quality of life?

Researchers will divide participants into two groups. One group will participate in the training program directly. The other group will first undergo a 12-week control intervention (i.e., standard treatment) before proceeding to the training program.

Participants will:

1. Take part in the individualized aerobic training program according to their baseline physical activity level for 12 weeks.
2. Visit the clinic once every 4 weeks for check-ups and tests.
3. Keep a diary of symptoms.

DETAILED DESCRIPTION:
This study is a single-center, semi-crossover, randomized controlled trial. Patients will be consecutively screened from gastroenterology and inflammatory bowel disease clinics. After obtaining informed consent, they are randomly assigned in a 1:1 ratio, stratified by diagnosis (CD and UC). Group A immediately begins a 12-week individualized exercise training program, while Group B starts with a 12-week control intervention, consisting only of routine diagnosis and treatment, followed by the 12-week individualized exercise training. Comparisons are made for all patients before and after the exercise training and the control intervention.

Participants will be given different progressive individualized aerobic training schedules based on their baseline physical activity levels, with the exercise intensity increased every 4 weeks.

The implementation of the training program is based on telemedicine, utilizing a combination of methods including wearable devices, WeChat groups, and online form submissions to ensure quality control over the duration, intensity, and quality of the exercise training. Participants are required to wear fitness bands during the exercise training and use exercise software to record the exercise process, including duration, trajectory, maximal heart rate, and average heart rate. These data are promptly sent to the researchers upon completion of the exercise. Before the commencement of the exercise program, a dedicated researcher instructs the participants on how to use the bands to record the type of exercise, duration, and maximum heart rate, and then to timely fill in the exercise records on the online forms. Additionally, the researchers will discuss with the participants at the outset about the individualized exercise (including location, frequency, intensity, and type), the participants' motivation, expectations, and goals, as well as potential difficulties, aiming to enhance adherence to the training program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CD or UC for more than 3 months.
* Disease activity in remission or mildly active (CD: CDAI < 220; UC: pMS < 5).
* Baseline physical activity intensity is low, measured by the IPAQ Chinese version short form, and without a habit of "regular exercise".
* Agree to participate in the study and accept a 12-week individualized aerobic exercise training program.

Exclusion Criteria:

* Pregnant or breastfeeding, or planning to become pregnant within the next 3 months.
* Presence of physical movement disorders or other chronic diseases that limit physical activity.
* Having an ileostomy.
* History of anal or intestinal surgery within the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (pVO2) (in ml/kg/min) | At baseline and the end of intervention at week 12
  Cardiorespiratory fitness measured by cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) | At baseline, week 4, week 8 and the end of intervention at week 12
  Measurement of patient-reported disease activity of CD participants. Higher scores mean higher activity. <150 indicates remission, 150~219 indicates mildly active.
Partial Mayo Score | At baseline, week 4, week 8 and the end of intervention at week 12
  Measurement of Patient-reported disease activity of UC participants. Higher scores mean higher activity. 0~1 indicates remission. 2~4 indicates mildly active.
Concentration of fecal calprotectin | At baseline and the end of intervention at week 12
Inflammatory Bowel Disease Questionnaire (IBDQ) | At baseline and the end of intervention at week 12
  32 questions grouped into four dimensions: bowel, systemic, social, and emotional. Scores range from 1 (poorest QoL) to 7 (best QoL). Higher scores indicate better QoL.
Fatigue severity scale (FSS) | At baseline and the end of intervention at week 12
  Minimum value is 9 and maximum value is 63 with higher scores indicating higher level of fatigue.
Hospital Anxiety and Depression Scale (HADS) | At baseline and the end of intervention at week 12
  Score of 0~21 with higher scores indicates higher level of anxiety and depression
International Physical Activity Questionnaire (IPAQ) short form | At baseline and the end of intervention at week 12
  A total IPAQ score is the sum of walking, moderate and vigorous metabolic equivalent of task (MET)-min/week.
Body Mass Index (BMI) in kg/m^2 | At baseline and the end of intervention at week 12
Waist circumference in cm | At baseline and the end of intervention at week 12
Concentration of serum fasting glucose in mmol/L | At baseline and the end of intervention at week 12
Concentration of serum albumin in g/L | At baseline and the end of intervention at week 12
Concentration of serum cholesterol in mmol/L | At baseline and the end of intervention at week 12
Concentration of serum triglyceride in mmol/L | At baseline and the end of intervention at week 12
Concentration of serum fasting lipoprotein in mmol/L | At baseline and the end of intervention at week 12
Concentration of serum uric acid in mmol/L | At baseline and the end of intervention at week 12
Oxygen uptake at aerobic threshold (in ml/kg/min) | at baseline and the end of intervention at week 12
  Oxygen uptake at aerobic threshold measured by CPET
Peak oxygen uptake per heart rate (in ml/kg/min) | at baseline and the end of intervention at week 12
  Peak oxygen uptake per heart rate measured by CPET
Maximal heart rate (in bpm) | At baseline and the end of intervention at week 12
  Maximal heart rate at peak measured by CPET
Six-Minute Walk Test (in meters) | At baseline and the end of intervention at week 12
  Maximum walked distance in meters conducted according to guideline
Exercise Benefits/Barriers Scale | At baseline and the end of intervention at week 12
  The Exercise Benefits/Barriers Scale (EBBS) will be used to assess participants' perceived benefits and barriers to exercise.
Plasma C-reactive protein (mg/L) | At baseline and end of the intervention at week 12
Plasma hemoglobin level (in g/L) | At baseline and end of the intervention at week 12
Body fat percentage (%) | At baseline and end of the intervention at week 12
  Body fat percentage measured via body composition analysis
Skeletal muscle mass (kg) | At baseline and end of the intervention at week 12
  Skeletal muscle mass (kg) measured via body composition analysis

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Lihuili Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start Date: Upon publication of this clinical trial. End Date: Five years following publication.
Access Criteria: Who can access the data? Researchers who provide a methodologically sound proposal.
  For what types of analysis? To achieve aims in the approved proposal. How can they access it? Proposals should be directed to drzhouying07@126.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Zhou Y, Liu H, Qian X, Zhang X, Xu F. Telemedicine-based individualised aerobic exercise training in Chinese adults with inactive or mildly active inflammatory bowel disease: study protocol for a single-centre, semi-crossover randomised controlled trial. BMJ Open. 2026 Jan 5;16(1):e103297. doi: 10.1136/bmjopen-2025-103297. PMID 41490862